CLINICAL TRIAL: NCT01104792
Title: Evaluation of the Long-term Safety, Tolerability, and Pharmacokinetics of Cariprazine in Patients With Schizophrenia
Brief Title: Long-term Study of Cariprazine in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGH-MD-11
Record Dates: First submitted 2010-04-12; First posted 2010-04-15 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Acute schizophrenia; Psychotropic drugs; Antipsychotic agents; Mental disorders; Dopamine agents; Central nervous system agents
MeSH Terms: conditions — Schizophrenia; Mental Disorders | interventions — cariprazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cariprazine (Experimental): Participants received cariprazine 3.0, 4.5, 6.0, or 9.0 mg orally once a day for 48 weeks.
  Interventions: Drug: Cariprazine

INTERVENTIONS:
Drug: Cariprazine — Cariprazine was supplied in capsules.
  Other Names: RGH-188

SUMMARY:
The objective of this study is to evaluate the long-term safety, tolerability, and pharmacokinetics of cariprazine in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients and corresponding caregivers who have provided informed consents prior to any study specific procedures.
* Patients currently meeting the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for schizophrenia (paranoid type, disorganized type, catatonic type, or undifferentiated type), as confirmed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (SCID).
* Patients with normal physical examination, laboratory, vital signs, and electrocardiogram (ECG).

Exclusion Criteria:

* Patients with a DSM-IV-TR diagnosis of schizoaffective disorder, schizophreniform disorder, bipolar I or bipolar II disorder, or psychotic disorders other than schizophrenia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 752 (Actual)
Dates: Start 2010-05-31 (Actual); Primary Completion 2013-01-31 (Actual); Study Completion 2013-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Migliore, MA, Study Director — Forest Laboratories
Locations (86):
- United States (39):
  - Forest Investigative Site 072, Little Rock, Arkansas
  - Forest Investigative Site 021, Little Rock, Arkansas
  - Forest Investigative Site 086, Little Rock, Arkansas
  - Forest Investigative Site 014, Springdale, Arkansas
  - Forest Investigative Site 080, Carson, California
  - Forest Investigative Site 079, Cerritos, California
  - Forest Investigative Site 048, Costa Mesa, California
  - Forest Investigative Site 070, Costa Mesa, California
  - Forest Investigative Site 022, Garden Grove, California
  - Forest Investigative Site 083, Garden Grove, California
  - Forest Investigative Site 050, Long Beach, California
  - Forest Investigative Site 006, Oceanside, California
  - Forest Investigative Site 003, Riverside, California
  - Forest Investigative Site 016, San Diego, California
  - Forest Investigative Site 073, Santa Ana, California
  - Forest Investigative Site 071, New Britain, Connecticut
  - Forest Investigative Site 002, Bradenton, Florida
  - Forest Investigative Site 041, Kissimmee, Florida
  - Forest Investigative Site 082, North Miami, Florida
  - Forest Investigative Site 055, Atlanta, Georgia
  - Forest Investigative Site 087, Atlanta, Georgia
  - Forest Investigative Site 012, Honolulu, Hawaii
  - Forest Investigative Site 018, Chicago, Illinois
  - Forest Investigative Site 008, Hoffman Estates, Illinois
  - Forest Investigative Site 044, Rockville, Maryland
  - Forest Investigative Site 007, Flowood, Mississippi
  - Forest Investigative Site 017, Creve Coeur, Missouri
  - Forest Investigative Site 076, Saint Charles, Missouri
  - Forest Investigative Site 045, St Louis, Missouri
  - Forest Investigative Site 052, Las Vegas, Nevada
  - Forest Investigative Site 004, Willingboro, New Jersey
  - Forest Investigative Site 040, Cedarhurst, New York
  - Forest Investigative Site 019, Willoughby, Ohio
  - Forest Investigative Site 077, Philadelphia, Pennsylvania
  - Forest Investigative Site 047, Philadelphia, Pennsylvania
  - Forest Investigative Site 074, Austin, Texas
  - Forest Investigative Site 084, DeSoto, Texas
  - Forest Investigative Site 043, Irving, Texas
  - Forest Investigative Site 078, Bellevue, Washington
- Colombia (4):
  - Forest Investigative Site 601, Bello, Antioquia
  - Forest Investigative Site 604, Pereira, Risaralda Department
  - Forest Investigative Site 602, Bogotá
  - Forest Investigative Site 605, Bogotá
- India (13):
  - Forest Investigative Site 503, Ahmedabad
  - Forest Investigative Site 519, Ahmedabad
  - Forest Investigative Site 501, Ahmedabad
  - Forest Investigative Site 500, Aurangabad
  - Forest Investigative Site 507, Kanpur
  - Forest Investigative Site 518, Lucknow
  - Forest Investigative Site 517, Mangalore
  - Forest Investigative Site 515, Mangalore
  - Forest Investigative Site 510, Mumbai
  - Forest Investigative Site 513, Nashik
  - Forest Investigative Site 509, Rajkot
  - Forest Investigative Site 506, Varanasi
  - Forest Investigative Site 505, Vijaywada
- Romania (6):
  - Forest Investigative Site 306, Bucharest
  - Forest Investigative Site 301, Cluj-Napoca
  - Forest Investigative Site 300, Craiova
  - Forest Investigative Site 311, Craiova
  - Forest Investigative Site 303, Târgovişte
  - Forest Investigative Site 304, Târgu Mureş
- Russia (12):
  - Forest Investigative Site 102, Arkhangelsk
  - Forest Investigative Site 103, Chelyabinsk
  - Forest Investigative Site 104, Chita
  - Forest Investigative Site 112, Saint Petersburg
  - Forest Investigative Site 105, Saint Petersburg
  - Forest Investigative Site 106, Saint Petersburg
  - Forest Investigative Site 113, Saint Petersburg
  - Forest Investigative Site 107, Saint Petersburg
  - Forest Investigative Site 109, Saint Petersburg
  - Forest Investigative Site 110, Saratov
  - Forest Investigative Site 108, Saratov
  - Forest Investigative Site 100, Tomsk
- Ukraine (12):
  - Forest Investigative Site 211, Hlevakha, Kyiv Oblast
  - Forest Investigative Site 206, Kherson, Stepanivka
  - Forest Investigative Site 208, Dnipropetrovsk
  - Forest Investigative Site 205, Dnipropetrovsk
  - Forest Investigative Site 200, Donetsk
  - Forest Investigative Site 203, Kharkiv
  - Forest Investigative Site 204, Kharkiv
  - Forest Investigative Site 201, Kyiv
  - Forest Investigative Site 202, Lviv
  - Forest Investigative Site 209, Poltava
  - Forest Investigative Site 210, Simferopol
  - Forest Investigative Site 207, Vinnytsia

REFERENCES:
- [Derived] Laszlovszky I, Barabassy A, Nemeth G. Cariprazine, A Broad-Spectrum Antipsychotic for the Treatment of Schizophrenia: Pharmacology, Efficacy, and Safety. Adv Ther. 2021 Jul;38(7):3652-3673. doi: 10.1007/s12325-021-01797-5. Epub 2021 Jun 6. PMID 34091867
- [Derived] Barabassy A, Sebe B, Acsai K, Laszlovszky I, Szatmari B, Earley WR, Nemeth G. Safety and Tolerability of Cariprazine in Patients with Schizophrenia: A Pooled Analysis of Eight Phase II/III Studies. Neuropsychiatr Dis Treat. 2021 Apr 7;17:957-970. doi: 10.2147/NDT.S301225. eCollection 2021. PMID 33854317
- [Derived] Nasrallah HA, Earley W, Cutler AJ, Wang Y, Lu K, Laszlovszky I, Nemeth G, Durgam S. The safety and tolerability of cariprazine in long-term treatment of schizophrenia: a post hoc pooled analysis. BMC Psychiatry. 2017 Aug 24;17(1):305. doi: 10.1186/s12888-017-1459-z. PMID 28836957

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The flexible-dose design for this study was selected to examine the relative safety and tolerability of a range of dosages of cariprazine. The starting dose of 1.5 mg/day was titrated as needed within the range of 3.0 - 9.0 mg/day based on the Investigator's judgment of response and tolerability.
Period: Overall Study
Arm/Group | Cariprazine
Started | 752
Completed | 226
Not Completed | 526
Not completed — Adverse Event | 77
Not completed — Insufficient Therapeutic Response | 22
Not completed — Protocol Violation | 45
Not completed — Withdrawal of Consent | 179
Not completed — Lost to Follow-up | 43
Not completed — Reasons Not Specified | 27
Not completed — Did Not Meet Eligibility Criteria | 133

BASELINE CHARACTERISTICS:
Population: The flexible-dose design for this study was selected to examine the relative safety and tolerability of a range of dosages of cariprazine. The starting dose of 1.5 mg/day was titrated as needed within the range of 3.0 - 9.0 mg/day based on the Investigator's judgment of response and tolerability.
Arm/Group | Cariprazine
Number analyzed (Participants) | 586
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178
  Male | 408
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48
  Not Hispanic or Latino | 523
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 68
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 229
  White | 250
  More than one race | 0
  Unknown or Not Reported | 35
Weight [Mean (Standard Deviation); unit: kg] | 79.94 (20.26)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.10 (5.80)
Waist circumference [Mean (Standard Deviation); unit: cm] — Summary statistics for this parameter based on 586 patients.
  cm | 91.76 (15.85)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 48 in the PANSS Total Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a 30-item rating scale that assesses the positive and negative symptoms of individuals with schizophrenia. Responses to the 30 items are based on a structured clinical interview with the patient and on supporting clinical information obtained from family, hospital staff, or other reliable informants. Of the 30 psychiatric parameters measured by the scale, 7 assess positive symptoms (eg, delusions, grandiosity); 7 assess negative symptoms (eg, blunted affect, emotional withdrawal); and 16 assess general psychopathology (eg, poor attention, active social avoidance). Each item is scored on a 7-point scale (1 = absent, 2 = minimal, 3 = mild, 4 = moderate, 5 = moderately severe, 6 = severe, and 7 = extreme). The PANSS total score can range from 30 to 210. A higher score indicates worse symptoms. A negative change score indicates improvement.
Time Frame: Baseline to Week 48
Population: Intent-to-treat population: All participants who took at least 1 dose of cariprazine and who had at least 1 post-baseline efficacy assessment. Only participants with data at both Baseline and Week 48 were included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cariprazine
Number analyzed (Participants) | 572
Units on a scale
  Baseline | 66.5 (12.1)
  Change From Baseline | -5.0 (14.0)

2. Secondary Outcome: Change From Baseline to Week 48 in the CGI-S Score
Description: The Clinical Global Impressions-Severity (CGI-S) scale is a 7-point scale that measures the overall severity of the illness compared with the severity of illness in other patients the Investigator has observed. The Investigator assesses the severity of the patient's illness as one of the following: 1 = Normal, not at all ill; 2 = Borderline ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; 7 = Among the most extremely ill patients. The CGI-S score can range from 1 to 7. A higher score indicates more severe illness. A negative change score indicates improvement.
Time Frame: Baseline to Week 48
Population: Intent-to-treat population: All participants who took at least 1 dose of cariprazine and who had at least 1 post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cariprazine
Number analyzed (Participants) | 578
Units on a scale
  Baseline | 3.0 (0.4)
  Change From Baseline | -0.1 (0.8)

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: The flexible-dose design for this study was selected to examine the relative safety and tolerability of a range of dosages of cariprazine. The starting dose of 1.5 mg/day was titrated as needed within the range of 3.0 - 9.0 mg/day based on the Investigator's judgment of response and tolerability.
  Safety population: All enrolled participants who took at least 1 dose of cariprazine.
Arm/Group | Cariprazine
All-Cause Mortality (participants affected / at risk) | 0/586
Serious Adverse Events (participants affected / at risk) | 59/586
Other Adverse Events (participants affected / at risk) | 419/586
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cariprazine (N=586)
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Medical device pain (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Cellulitis (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Gun shot wound (Injury, poisoning and procedural complications) | 1
Muscle injury (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Brain injury (Nervous system disorders) | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Schizophrenia (Psychiatric disorders) | 25
Psychotic disorder (Psychiatric disorders) | 12
Suicidal ideation (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 2
Hallucination, auditory (Psychiatric disorders) | 2
Schizophrenia, paranoid type (Psychiatric disorders) | 2
Aggression (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 1
Homicidal ideation (Psychiatric disorders) | 1
Paranoia (Psychiatric disorders) | 1
Psychotic behaviour (Psychiatric disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/178
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Social stay hospitalisation (Social circumstances) | 6
Hospitalisation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cariprazine (N=586)
Nausea (Gastrointestinal disorders) | 51
Dyspepsia (Gastrointestinal disorders) | 42
Constipation (Gastrointestinal disorders) | 33
Toothache (Gastrointestinal disorders) | 31
Diarrhoea (Gastrointestinal disorders) | 30
Nasopharyngitis (Infections and infestations) | 30
Weight increased (Investigations) | 79
Blood creatine phosphokinase increased (Investigations) | 35
Akathisia (Nervous system disorders) | 118
Headache (Nervous system disorders) | 104
Extrapyramidal disorder (Nervous system disorders) | 47
Tremor (Nervous system disorders) | 46
Dizziness (Nervous system disorders) | 32
Insomnia (Psychiatric disorders) | 104
Anxiety (Psychiatric disorders) | 68
Restlessness (Psychiatric disorders) | 49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.